CLINICAL TRIAL: NCT00032019
Title: Phase II Study Of Dose-Adjusted Epoch-Rituximab (EPOCH-R) Chemotherapy For Patients With Previously Untreated Aggressive CD20+ B-Cell Non-Hodgkin's Lymphoma (NHL)
Brief Title: Combination Chemotherapy and Monoclonal Antibody Therapy in Treating Patients With Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-50103; U10CA031946 (NIH); CALGB-50103; CDR0000069249 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Lymphoma
Keywords: stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Rituximab; Cyclophosphamide; Doxorubicin; Etoposide; Prednisone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EPOCH-Rituximab (Experimental): Addition of monoclonal antibody therapy to chemotherapy for treatment of pts with aggressive CD20+ NHL
  Interventions: Biological: filgrastim; Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: prednisone; Drug: vincristine sulfate

INTERVENTIONS:
Biological: filgrastim — Cycle 1: 300 ug (BW < = 70 kg) or 480ug (BW >70 kg) sub Q injection Day 6 until ANC > 5000/uL after nadir counts Subsequent cycle dosages based on previous cycle toxicity or Day 1 Tx toxicity
  Other Names: G-CSF
Biological: rituximab — 375 mg/sq m IV infusion Day 1 Cycle 1 Subsequent cycle dosage based on previous cycle or day 1 of tx toxicities
Drug: cyclophosphamide — 750 mg/sq m IV infusion on Day 5 Cycle 1 Subsequent cycle dosage based on previous cycle or day 1 treatment toxicities
Drug: doxorubicin hydrochloride — 10 mg/sq m/day continuous IV infusion on Days 1-4 Cycle 1 Subsequent cycle dosages based on previous cycle and Day 1 treatment toxicities
Drug: etoposide — 50 mg/sq m/day continuous IV infusion Days 1-4 Cycle 1 Subsequent cycle dosages based on previous cycle and day 1 of treatment toxicities
Drug: prednisone — 60 mg/sq m PO bid days 1-5 of ea cycle
Drug: vincristine sulfate — 0.4 mg/sq m/day continuous IV infusion uncapped on Days 1-4 Cycle 1 Subsequent cycle dosages based on previous cycle and day 1 of treatment toxicities

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies such as rituximab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Combining rituximab with combination chemotherapy may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combining rituximab with combination chemotherapy in treating patients who have previously untreated non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate, progression-free survival, and overall survival of patients with previously untreated aggressive CD20+ B-cell diffuse large cell or immunoblastic large cell lymphoma treated with rituximab, doxorubicin, etoposide, vincristine, prednisone, and cyclophosphamide.
* Determine the toxic effects of this regimen in these patients.
* Correlate tumor proliferation rate (MIB-1), bcl-2 expression, and p53 overexpression with complete response rate, progression-free survival, and overall survival in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive rituximab IV on day 1; doxorubicin IV continuously, etoposide IV continuously, and vincristine IV continuously on days 1-4; oral prednisone twice daily on days 1-5; and cyclophosphamide IV on day 5. Patients also receive filgrastim (G-CSF) subcutaneously beginning on day 6 and continuing until blood counts recover. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity. After 4 courses, patients with complete or partial response receive 2 additional courses.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 25-50 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage II, III, or IV diffuse large cell lymphoma and WHO variants

  * CD20+ large B-cell lymphoma, including those with immunoblastic features
  * CD20+ thymic B-cell lymphoma
  * No evidence of indolent lymphoma
  * No mantle cell lymphomas or equivocal B-cell lymphomas that express markers of mantle cell lymphoma (e.g., cyclin D) or other subtypes
* No known lymphomatous involvement of the CNS, including the parenchyma or leptomeninges

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* CALGB 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,000/mm3*
* Platelet count at least 100,000/mm3* NOTE: * Unless due to lymphoma

Hepatic:

* Bilirubin no greater than 2.0 mg/dL* NOTE: * Unless due to lymphoma or Gilbert's disease

Renal:

* Creatinine no greater than 1.5 mg/dL* NOTE: * Unless due to lymphoma

Cardiovascular:

* LVEF greater than 45%
* No ischemic heart disease
* No myocardial infarction or congestive heart failure within the past year

Other:

* HIV negative
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior cytotoxic chemotherapy
* No other concurrent chemotherapy

Endocrine therapy:

* Prior short-course of glucocorticoids allowed
* No concurrent hormones except for non-disease-related conditions (e.g., insulin for diabetes)
* No concurrent steroids except for adrenal failure
* No concurrent dexamethasone or other steroidal antiemetics

Radiotherapy:

* Prior limited-field radiotherapy allowed

Surgery:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2002-02; Primary Completion 2004-12 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Response | 5 months

SECONDARY OUTCOMES:
Progression free Survival | Study entry to progression or tx related death
Overall survival | Study entry to death from any cause
Toxicity | q 2cycles on Tx, then q 6 mon for 2 yrs, then at relapse

CONTACTS AND LOCATIONS:
Overall Officials: Wyndham H. Wilson, MD, PhD, Study Chair — National Cancer Institute (NCI)
Locations (81):
- United States (80):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Cedars-Sinai Comprehensive Cancer Center at Cedars-Sinai Medical Center, Los Angeles, California
  - Naval Medical Center - San Diego, San Diego, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Memorial Regional Hospital Comprehensive Cancer Center, Hollywood, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Saint Anthony Medical Center, Rockford, Illinois
  - Fort Wayne Medical Oncology and Hematology, Incorporated, Fort Wayne, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Baptist Hospital East - Louisville, Louisville, Kentucky
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Lakeland Cancer Care Center at Lakeland Hospital - St. Joseph, Saint Joseph, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - Las Vegas, Las Vegas, Nevada
  - New Hampshire Oncology-Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth Medical School, Lebanon, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., East Syracuse, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - University Hospital at State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Veterans Affairs Medical Center - Asheville, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - NorthEast Oncology Associates, Concord, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - Lenoir Memorial Hospital Cancer Center, Kinston, North Carolina
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Oklahoma University Medical Center at University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Lifespan: The Miriam Hospital, Providence, Rhode Island
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Green Mountain Oncology Group, Bennington, Vermont
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Virginia Oncology Associates - Norfolk, Norfolk, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., Roanoke, Virginia
  - St. Mary's Medical Center, Huntington, West Virginia
- Puerto Rico Cancer Center at University of Puerto Rico - Medical Sciences Campus, San Juan, Puerto Rico

REFERENCES:
- [Result] Hsi ED, Said J, Johnson JL, et al.: Biologic prognostic markers in diffuse large B-cell lymphoma patients treated with dose adjusted EPOCH-R: a CALGB 50103 correlative science study. [Abstract] Blood 112 (11): A-476, 2008.
- [Result] Wilson WH, Porcu P, Hurd D, et al.: Phase II study of dose-adjusted EPOCH-R in untreated de novo CD20+ diffuse large B-cell lymphoma (DLBCL)-CALGB 50103. [Abstract] J Clin Oncol 23 (Suppl 16): A-6530, 567s, 2005.
- [Derived] Wilson WH, Jung SH, Porcu P, Hurd D, Johnson J, Martin SE, Czuczman M, Lai R, Said J, Chadburn A, Jones D, Dunleavy K, Canellos G, Zelenetz AD, Cheson BD, Hsi ED; Cancer Leukemia Group B. A Cancer and Leukemia Group B multi-center study of DA-EPOCH-rituximab in untreated diffuse large B-cell lymphoma with analysis of outcome by molecular subtype. Haematologica. 2012 May;97(5):758-65. doi: 10.3324/haematol.2011.056531. Epub 2011 Dec 1. PMID 22133772